CLINICAL TRIAL: NCT04826198
Title: An Open-label, Multicentric, Phase Ib/II Study to Assess the Safety and Efficacy of AsiDNATM, a DNA Repair Inhibitor, Administered Intravenously in Addition to Niraparib in Patients With Relapsed Platinum Sensitive Ovarian Cancer Already Treated With Niraparib Since at Least 6 Months
Brief Title: Safety and Efficacy of AsiDNATM, a DNA Repair Inhibitor, Administered Intravenously in Addition to PARP Inhibitors in Patients With Relapsed Platinum Sensitive Ovarian Cancer Already Treated With PARP Inhibitors Since at Least 6 Months
Acronym: REVOCAN
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Treatment availability issue: The manufacturer of AsiDNA™ decided to cease production to develop an improved version, and the contract ensuring access to this molecule has expired.
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-000825-18; 2020-3047 (Other: CSET number)
Record Dates: First submitted 2021-02-23; First posted 2021-04-01 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — niraparib; olaparib; rucaparib

STUDY DESIGN:
Intervention Model Description: Multicenter, open label, phase Ib/II
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AsiDNA in addition to Niraparib (Experimental): Part A: AsiDN in addition to Niraparib (Safety evaluation) Part B: AsiDN in addition to Niraparib (Efficacy evaluation and Safety confirmation )
  Interventions: Drug: AsiDNA; Drug: Niraparib; Drug: Olaparib; Drug: Rucaparib

INTERVENTIONS:
Drug: AsiDNA — Unit dose: Vial containing 100 mg of AsiDNA™ (free acid) Regimen: 3 consecutive infusions (D1, D2, D3) followed by a once a week iv infusion on D8 and D15 of a 21 day-treatment cycle at first cycle, then weekly iv infusion in the absence of disease progression or unacceptable toxicity Mode/route: 1 hour intravenous (iv) infusion
Drug: Niraparib — Unit dose: Hard capsule containing 100mg of Niraparib Regimen: The last dose given during the 6 previous months of Niraparib 200 mg/day or 300 mg/day, (or 100 mg/day only if the patient has received this dose since at least 6 months) Daily, 1, 2 or 3 hard capsules at 100mg once daily at approximately the same time each day.
  Mode/route: Per os
Drug: Olaparib — Product name: Olaparib Pharmaceutical form: Tablets containing 100 or 150mg of Olaparib Route of administration: per os Dose Regimen: The last dose given during the 6 previous months of Olaparib 600 mg/day or 500 mg/day, (or 400 mg/day only if the patient has received this dose since at least 6 months) Two times daily (300mg or 250 mg or 200mg) at approximately the same time each day.
Drug: Rucaparib — Product name: Rucaparib Pharmaceutical form: Tablets containing 200 or 250 or 300mg of Rucaparib Route of administration: per os Dose Regimen: The last dose given during the 6 previous months of Rucaparib 1200 mg/day or 1000 mg/day, or 800mg/day (or 600 mg/day only if the patient has received this dose since at least 6 months) Two times daily (600mg or 500mg or 400mg or 300mg) at approximately the same time each day.

SUMMARY:
The objective of REVOCAN study is to assess the abrogation of PARP inhibitors resistance in patients with relapsed platinum sensitive ovarian cancer treated with PARP inhibitors in maintenance since at least 6 months and who have only an increase of CA 125 without any progression according to RECIST criteria. AsiDNATM at 600 mg will be tested in addition to PARP inhibitors given according to the label in REVOCAN study.

ELIGIBILITY:
Inclusion Criteria:

1. Patient should understand, sign, and date the written informed consent form prior to any protocol-specific procedures performed. Patient should be able and willing to comply with study visits and procedures as per protocol.
2. Female aged ≥ 18 years (no upper limit of age) at the time of consent signature.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
4. Life expectancy of at least 3 months.
5. Histologically diagnosed ovarian cancer, fallopian tube cancer or primary peritoneal cancer regardless BRCA status.
6. Availability of BRCA status;
7. Patient has received at least 2 previous courses of platinum-containing therapy and has a disease that was considered platinum sensitive that means in response (complete or partial) to the last platinum course leading to the administration of Niraparib, or Rucaparib, or Olaparib (PARP inhibitors).
8. The patient has received Niraparib in maintenance for at least 6 months and who has only an increase of CA125 at least twice the upper limit of normal within 2 weeks prior to starting treatment without any progression according to RECIST criteria or according to clinical assessment
9. Patient should be treated within 2 weeks after CT scan without any progression according to RECIST criteria
10. Patient with adequate biological parameters at baseline defined as:

    * absolute neutrophil count (ANC) ≥ 1.5 x 109/L,
    * hemoglobin (Hb) level ≥ 9g/dL,
    * platelet count ≥ 100 x 109/L,
    * total bilirubin level ≤ 1.5 Upper Limit Normal (ULN),
    * aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 2.5x ULN
    * calculated glomerular filtration rate (GFR) ≥ 60 mL/min/1.73m2 (per Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula),
    * INR ≤ 1.2 (except if patient treated with anti-vitamine K); anticoagulation with anti-vitamin K and Low Molecular Weight Heparin [LMWH] is allowed.
11. Patient of childbearing potential must agree to use adequate contraception prior to study entry, during the study and for 3 months after the study participation
12. Patient of childbearing potential must have a serum negative pregnancy test within 4 days prior to first administration. Females who are postmenopausal for at least 1 year (defined as more than 12 months since last menses) or are surgically sterilized do not require this test.
13. Patient must be affiliated to a social security system or an equivalent system.

Exclusion Criteria:

1. Patient has mucinous or clear cell subtypes of epithelial ovarian cancer, carcinosarcoma or undifferentiated ovarian cancer
2. Patient treated concomitantly with bevacizumab
3. Patient previously treated with PARPi as first line maintenance
4. Other Malignancy within the last 5 years except curatively treated nonmelanoma skin cancer or in situ carcinoma of the cervix, and in situ breast cancer
5. Patient with central nervous system (CNS) metastases;
6. Other tumor location necessitating an urgent therapeutic intervention (e.g., palliative care, surgery or radiation therapy, such as spinal cord compression, other compressive mass, uncontrolled painful lesion, bone fracture).
7. Patient with uncontrolled disease-related metabolic disorder (e.g., hypercalcemia, SIADH) or uncontrolled diabetes.
8. Quantitative total urine protein > 1.0 g/24 hour at baseline
9. Patient with uncontrolled congestive heart failure defined as New York Heart Association (NYHA) class III or IV, uncontrolled hypertension, unstable heart disease (e.g., coronary artery disease with unstable angina or myocardial infarction within 6 months before study treatment administration).
10. Patient with significant ECG abnormalities defined as any cardiac dysrhythmia (> grade 2) (i.e., significant ventricular arrhythmia as persistent ventricular tachycardia and/or ventricular fibrillation; severe conduction disorders as atrio-ventricular block 2 and 3, sino-atrial block) or baseline QT/QTc interval >480 milliseconds (ms).
11. Patient with significant chronic liver disease (e.g., significant fibrosis,known cirrhosis) or active HBV or HCV infection; if AgHbs positive, an effective antiviral treatment to prevent hepatitis B reactivation is recommended.
12. Patient with HIV infection or an active infection requiring specific antiinfective therapy are not eligible until all signs of infection have resolved, and this within 2 weeks prior to the first study treatment administration.
13. Patient whose medical, psychological including alcohol or drug abuse, or surgical conditions are unstable and may affect the study completion and/or compliance and/or the ability to give informed consent.
14. Participation in another clinical trial with any investigational drug within 28 days prior to first study drug administration.
15. Vulnerable adult patients benefiting from a specific legal protection status.
16. Patient who has received mouse antibodies (unless the assay used has been shown not to be influenced by HAMA4,5) or if there has been medical and/or surgical interference with their peritoneum or pleura during previous 28 days
17. Patient pregnant or breastfeeding

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Ovarian cancer
Enrollment: 13 (Actual)
Dates: Start 2020-10-05 (Actual); Primary Completion 2024-04-04 (Actual); Study Completion 2024-04-04 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicities (DLT) | 21 days
  Occurrence of cases of Dose Limiting Toxicity (DLT) will be recorded and reviewed according to a predefined definition.
  DLTs include the following specific treatment-related AEs occurring during the first 21 days (from D1 to D21) treatment period (based on the National Cancer
  Institute [NCI] Common Terminology Criteria for Adverse Events (AE) [CTCAE] scale, version 5.0 defined as:
  * Haematological toxicity:
    1. Grade 4 neutropenia lasting ≥ 7 days,
    2. Febrile Neutropenia,
    3. Grade 4 thrombocytopenia or grade 3 thrombocytopenia associated with bleeding.
  * Non haematological toxicity:
  Any drug-related non-hematological toxicity grade ≥ 3 toxicity (except alopecia, fatigue, nausea, controlled hypertension and vomiting adequately treated with antiemetic treatment and non-clinically significant laboratory values abnormalities).

CONTACTS AND LOCATIONS:
Locations (6):
- France (6):
  - CHU Jean Minjoz, Besançon, Besancon
  - Hospices civils de Lyon(CHU Lyon Sud), Pierre-Bénite, Lyon
  - Institut de Cancérologie de l'Ouest - St Herblain, Saint-Herblain, Nantes
  - Gustave Roussy, Villejuif, Val De Marne
  - Institut Bergonié, Bordeaux
  - Centre Antoine Lacassagne, Nice

IPD SHARING:
Plan to Share IPD: Undecided